CLINICAL TRIAL: NCT00453700
Title: Prevalence of Chagas Disease in Immigrant Patients With Conduction Abnormalities on Electrocardiogram
Status: Completed | Type: Observational
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sheba Meymandi, Principal Investigator, University of California, Los Angeles
Other Study IDs: 06H-561004
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2007-03

CONDITIONS: Chagas Disease
Keywords: chagas; trypanosoma cruzi
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- serological testing: In Latin American immigrants diagnosed with nonischemic cardiomyopathy in Los Angeles, serological testing for Trypanosoma cruzi was performed at enrollment.
  Interventions: Procedure: Trypanosoma cruzi serology

INTERVENTIONS:
Procedure: Trypanosoma cruzi serology

SUMMARY:
Chagas disease is endemic to the Americas, infecting between 16-18 million individuals. In immigrant populations in the United States from endemic areas, it is estimated up to 4.9% may be asymptomatic carriers of Trypanosoma cruzi, the organism which causes Chagas disease. Between 10-20% of these patients progress to development of end-stage cardiomyopathy with a high associated morbidity. Following acute disease, patients enter into an indeterminate phase which can last 10-20 years. The earliest sign of cardiac involvement usually is electrocardiogram abnormalities. The most common abnormality is right bundle branch block (RBBB), followed by left anterior fascicular block (LAFB), and left bundle branch block (LBBB). Recent studies have shown that treatment of patients at this stage with antiparasitics may delay the progression of overt cardiomyopathy.

At the University of California, Los Angeles, there is a large population of immigrant patients from countries endemic to Chagas disease. The researchers propose that screening patients with conduction abnormalities on electrocardiogram may be a potentially useful method to identify patients with early cardiac manifestations of Chagas disease. The researchers hope to enroll approximately 300 individuals with RBBB, LAFB or LBBB on electrocardiogram to determine the incidence of Chagas disease in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* One of the following EKG abnormalities:

  * Complete or incomplete right bundle branch block (RBBB)
  * Left anterior fascicular block (LAFB)
  * Left bundle branch block (LBBB)
* Residence at any point in past in an endemic area (any country in Central or South America or Mexico) for at least 12 months.
* Age >18 and <60.

Exclusion Criteria:

* Ejection fraction <40%
* Symptomatic heart failure
* Documented coronary artery disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All Latin American immigrant patients with newly diagnosed nonischemic cardiomyopathy at one U.S. medical center were asked to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of positive trypanosoma cruzi serologies | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sheba K Meymandi, M.D., Principal Investigator — OV-UCLA Medical Center
Locations (1):
- OV-UCLA Medical Center, Sylmar, California, United States